CLINICAL TRIAL: NCT06950749
Title: Effects of Robotic Gloves Along With Task-oriented Mirror Therapy on Motor Functions of Hands in Sub-acute Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/50
Record Dates: First submitted 2024-11-14; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Mirror Therapy; Robotics; Neurorehabilitation
Keywords: stroke; mirror therapy; robotics; neurorehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTERVENTION GROUP (A) (Experimental): INTERVENTION GROUP (A) will receive Robotic Gloves Assisted Task-Oriented Mirror Therapy along with conventional therapy.
  subjects will sit on a chair and placed their both hands on the table. Patients will wear the soft robotic glove on affected hand and the data glove the unaffected hand.
  Subjects will be instructed to visually observe the hand being moved by soft robotic glove
  * In mirror training mode: Synchronized flexion and extension training with both hands.
  * Task oriented activities: With help of robot patient will practice grasping, releasing the tennis ball, positioning the cup upright, carrying a wooded block, putting a ball
  Interventions: Procedure: Robotic Gloves assisted Task-oriented mirror therapy
- INTERVENTIONAL GROUP (B) (Experimental): INTERVENTIONAL GROUP (B) will receive Task-Oriented Mirror Therapy along with conventional therapy.
  Both the extremities of the subject will be placed on the table and mirror will be placed in the patients' mid sagittal plane. Mirror will be placed in such a way that the reflection of the non-affected arm to be seen.
  * Grasping and releasing (cylindrical grasp, spherical grasp, hook grasp, pincer grasp)
  * Task oriented activities: positioning the cup upright, carrying a wooded block and putting a ball.
  Interventions: Procedure: Task-Oriented Mirror Therapy

INTERVENTIONS:
Procedure: Robotic Gloves assisted Task-oriented mirror therapy — Robotic gloves assissted task-oriented Mirror therapy along with conventional therapy.
  Conventional therapy consists of stretching exercises,active assisted and active ROMS of shoulder along with weight bearing and reaching activities.
  Robotic gloves assisted task-oriented Mirror therapy will be delivered by syrebo robotic hand rehabilitation device.
  it has different training modes including Mirror mode and task-oriented training.
  5 sessions per week will be provided for 8 weeks exercises: 30 minutes (3 sets of 10 reps)
  * In mirror training mode: Synchronized flexion and extension training with both hands.
  Arms: INTERVENTION GROUP (A)
Procedure: Task-Oriented Mirror Therapy — Interventional group (B) will receive Task-Oriented Mirror Therapy along with conventional therapy.
  To perform Task-Oriented Mirror Therapy both the extremities of the subject will be placed on the table and the mirror (40×60 cm) will be placed in the patients' mid-sagittal plane. Mirror will be placed in such a way that the reflection of the non-affected arm can be seen. The subjects will be instructed to perform the movement bilaterally. The movement on the impaired limb will be performed. Affected arm is involved in exercise therapy either through patients trying to move themselves or with a therapist in assisting movement.
  5 sessions per week will be provided for 8 weeks.
  * Task-Oriented Mirror therapy exercises: 30 minutes. (3 sets of 10 reps)
  * Hand flexion and extension through the tennis ball.
  * Grasping and releasing (cylindrical grasp, spherical grasp, hook grasp, pincer grasp)
  * Task oriented activities: positioning the cup upright, carrying a woode
  Arms: INTERVENTIONAL GROUP (B)

SUMMARY:
This study is randomized control trial and purpose of this study is to find effects of robotic gloves assisted task-oriented mirror therapy in comparison with task-oriented mirror therapy on motor functions of hand in sub-acute stroke patients.

DETAILED DESCRIPTION:
Motor functions of the hand involve different movements and activities that the hand can perform due to the coordination of different muscles group in everyday activities which involves dexterity, manipulative skills and task performance skills which includes grasp, release and different types of grips of hand.

RATIONALE:

While the mirror therapy has been studied extensively and literature provide good quality of evidence for effects of mirror therapy on motor functions of hands the integration of pneumatic Robotic Mirror Therapy is relatively less explored .

and there is no comparison between Task oriented MT and pneumatic Robotic Mirror Therapy

SIGNIFICANCE This study will increase the understanding and therapeutic potential of robotic gloves assisted task-oriented MT mirror therapy and will demonstrate its efficacy as beneficial interventions.

Modern devices like robotic gloves can potentially increase patient compliance by providing positive outcomes, setting goals and improving functional performance.

They can make therapy more engaging, interactive and help the patients track their progress, which can motivate them to adhere to their rehabilitation program.

HYPOTHESIS ALTERNATE HYPOTHESIS There will be a statistically significant difference in the effects of Task oriented Mirror Therapy in comparison with Robotic gloves Assisted task-oriented Mirror Therapy on motor functions of hand in patients with sub-acute Stroke (p<0.05).

NULL HYPOTHESIS There will be no statistically significant difference in the effects of Task oriented Mirror Therapy in comparison with Robotic gloves Assisted task-oriented Mirror Therapy on motor functions of hand in patients with sub-acute Stroke (p>0.05).

ELIGIBILITY:
Inclusion Criteria:

* 40 years and above.
* Ischemic (MCA) stroke.
* Male and females both.
* Montreal Cognitive Assessment (MoCA score >24 points).
* Motor power of proximal upper Extremity at least 3 with ability to reach out.
* FMA score for upper Extremity below 47
* Modified Ashworth spasticity score <2 in hands and finger joints.
* Ability to sit for at least 60 minutes

Exclusion Criteria:

* Musculoskeletal problems such as severe pain in any joints of the paretic upper extremity.
* Contractures in shoulder, elbow, hand or finger joints.
* Severe Visual impairments.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
hand motor functions | 08 Weeks
  Fugl Meyer Assessment (FMA-UE), wii be used to assess motor functions of hands FMA:used to measure motor recovery in stroke patients. it has a maximum score of 66 points FMA hand section will be used to assess motor functions of hands from baseline to end of interventions.
Dexterity | 8 weeks
  An action research arm test will be used. Scores were rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally) for a maximum score of 57.
unilateral gross manual dexterity | 8 weeks
  Box and block test is used to assess the unilateral gross manual dexterity of the hand. Subjects will be asked to move a wooden block from one compartment to the other.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan